CLINICAL TRIAL: NCT04871477
Title: The Adoption of Audio Recording in the Outpatient Supportive Care Center
Brief Title: Adoption of Audio Recording in the Outpatient Supportive Care Center
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0240; NCI-2021-02621 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0240 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-05; First posted 2021-05-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (audio recording): Patients audio record the recommendations and instructions given to them by the doctor record as part of their clinic visit at the Supportive Care Center.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Audio record part of clinic visit
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study evaluates how patients feel about having an audio recording of their visit to help remember information given to them and share that information with family members and/or caregivers not present during a clinic visit. Information from this study may help evaluate the effectiveness of using technology to help improve patient care by recording consultation recommendations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the patient's perception of the usefulness of the audio recording in helping to recall information given to him/her in the visit along with the perception of usefulness in the dissemination of information to family member(s) and/or caregiver(s) not present at the clinic visit.

SECONDARY OBJECTIVES:

I. To assess the number of times the recording is listened to. II. To assess the ease of use of the technology. III. To assess the ability to share the information with the patient's family member(s) and/or caregiver(s) if he or she chooses to do so.

IV. To assess the patient perception of whether the audio recording caused any disruption to the clinic.

V. To estimate the participation rate of patients. VI. To explore association between patient's perception of the usefulness of the audio recording and patient's demographic/clinical characteristics.

VII. To explore the association between age and sex of the caregiver and frequency of caregiver's use of the audio recording.

VIII. To explore the association of the ease of use of the technology and the type of device and application used.

OUTLINE:

Patients audio record the recommendations and instructions given to them by the doctor record as part of their clinic visit at the Supportive Care Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of advanced cancer as defined as locally advanced, recurrent or metastatic cancer. Both solid and liquid tumors are eligible for the study
* Patients who are seen in the outpatient supportive care center at M.D. Anderson Cancer Center
* Patients who have access to a recording device or cellphone with recording technology
* Patients who can be contacted 7 to 11 days from the clinic visit that the recording took place
* Patients who can sign informed consent
* Patients who are able to read and write in English
* Patients 18 years or older

Exclusion Criteria:

* Patients who have been diagnosed with delirium or cognitive impairment. This will be defined by chart review along with review of the MD Anderson Symptom Inventory (MDAS) the day of clinic visit. An MDAS of 7 or greater will be considered to define delirium in this study
* Patients who are unwilling to sign informed consent
* Patients who have used audio recordings before in clinic visits
* Patients who have severe hearing impairments without access to assisted devices or programs to aid in listening to the recorded material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who will select "Complete Agree/Partially Agree" in Question 1 "I found the audio recording useful after the visit" | through study completion, an average of 1 year
  Will be summarized using proportion along with a 95% confidence interval.
Proportion of patients who will select "Complete Agree/Partially Agree" in Question 2 "I was able to effectively discuss my medical condition with my family member(s) and/or caregiver(s) who were not present at the clinical visit | through study completion, an average of 1 year
  Will be summarized using proportion along with a 95% confidence interval.

SECONDARY OUTCOMES:
Number of times the recording is listened to | through study completion, an average of 1 year
  Descriptive statistics will be used to summarize the results. Wilcoxon rank sum test or Kruskal-Wallis test will be applied to examine differences in continuous variables between or among patient's demographic/clinical characteristics.
To assess the ease of use of the technology. | through study completion, an average of 1 year
  Descriptive statistics will be used to summarize the results. Chi squared test or Fisher's exact test will be applied to examine the association between the ease of use of the technology and patient's demographic/clinical characteristics.
To assess the ability to share the information with the patient's family member(s) and/or caregiver(s) if he or she chooses to do so. | through study completion, an average of 1 year
  Descriptive statistics will be used to summarize the results. Chi-squared test or Fisher's exact test will be applied to examine the association between the ability to share and patient's demographic/clinical characteristics.
To assess the patient perception of whether the audio recording caused any disruption to the clinic | through study completion, an average of 1 year
  Descriptive statistics will be used to summarize the results. Chi-squared test or Fisher's exact test will be applied to examine the association between the patient perception of whether audio recording caused any disruption to the clinic and patient's demographic/clinical characteristics.
Patient participation rate | through study completion, an average of 1 year
  The participation rate of patients in this study will be estimate using proportion along with 95% confidence interval.
To explore the association between the frequency of caregivers' use of audio recording | through study completion, an average of 1 year
  Pearson or Spearman correlation coefficient will be used to assess the association between caregivers' age and frequency of their use of the audio recording. Wilcoxon rank sum test will be applied to examine differences in frequency of caregivers' use of audio recording between their sexes.
To explore the association of the ease of use of the technology and the type of device and application used | through study completion, an average of 1 year
  Chi-squared test or Fisher's exact test will be applied to examine the association between the ease of use of the technology and the types of recording devices/applications.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States